CLINICAL TRIAL: NCT03531229
Title: Interventional, Randomized, Double-blind, Sequential-group, Placebo-controlled, Single-ascending-oral-dose Study Investigating the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of Lu AF76432 in Healthy Young Men
Brief Title: Single Ascending Dose Study of Lu AF76432 in Healthy Young Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 17479A
Record Dates: First submitted 2018-04-20; First posted 2018-05-21 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: 36 Subjects are planned for enrolment, with 6 subjects per cohort. The subjects will be randomized to Lu AF76432 or placebo in a 4:2 ratio per cohort. A maximum of 2 additional cohorts of young healthy men will be permitted thereby allowing investigation of a maximum of 48 subjects
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo to Lu AF76432
  Interventions: Drug: Placebo
- Lu AF76432 (Experimental): Lu AF76432
  Interventions: Drug: Lu AF76432

INTERVENTIONS:
Drug: Placebo — Placebo to Lu AF76432 oral solution
  Arms: Placebo
Drug: Lu AF76432 — Lu AF76432 oral solution 2.5 mg/ml. Starting dose will be 3,5 mg, actual doses for following cohorts will be defined based on results from preceding dosing group(s).
  Arms: Lu AF76432

SUMMARY:
The purpose of this study is to investigate safety, tolerability and pharmacokinetics of the drug Lu AF76432 given as single oral ascending doses to healthy young men

ELIGIBILITY:
Inclusion Criteria:

-Healthy young non-smoking men ≥18 years of age and ≤45 years of age at the Screening Visit and a body mass index (BMI) ≥18.5kg/m2 and ≤30kg/m2 at the Screening Visit.

Exclusion Criteria:

* The subject has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder or the subject is, in the opinion of the investigator, unlikely to comply with the protocol or is unsuitable for any reason
* The subject has taken any investigational medicinal product <3 months prior to the first dose of IMP

Other inclusion and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events | From dosing to 12 days
  Safety and Tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, weight, ECG parameters and physical examination)

SECONDARY OUTCOMES:
AUC0-t | From dosing to 72 hours post dose
  Area under the plasma concentration-time curve from zero to time t
Cmax | From dosing to 72 hours post dose
  Maximum observed concentration
AUC0-inf | From dosing to 72 hours post dose
  Area under the plasma concentration-time curve from zero to infinity
CL/F | From dosing to 72 hours post dose
  Oral clearance

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Parexel Early Phase Clinical Unit, Harrow, United Kingdom